CLINICAL TRIAL: NCT05198817
Title: A Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of SHR-2002 Injection or in Combination With Other Anti-cancer Therapy in Advanced Malignant Tumors of Patients
Brief Title: A Trial of SHR-2002 Injection or Combined With Other Anti-cancer Medication in Advanced Malignant Tumors of Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2002-I-101
Record Dates: First submitted 2022-01-03; First posted 2022-01-20 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — Injections; SHR-1701

STUDY DESIGN:
Intervention Model Description: SHR-2002 injection monotherapy and in combination with other anti-cancer therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: SHR-2002 injection、Camrelizumab for Injection, SHR-1316 injection, SHR-1701 injection

INTERVENTIONS:
Drug: SHR-2002 injection、Camrelizumab for Injection, SHR-1316 injection, SHR-1701 injection — Firstly Dose Escalation and Dose Expansion of SHR-2002 injection monotherapy should be conducted. After RP2D and MTD of the SHR-2002 injection monotherapy were confirmed, Dose Escalation, Dose Expansion and Efficacy Expansion of SHR-2002 injection in combination with other anti-cancer treatment would be completed, including Camrelizumab for Injection, or SHR-1316 injection, or SHR-1701 injection.

SUMMARY:
The study is being conducted to evaluate safety, tolerability, pharmacokinetics and preliminary efficacy of SHR-2002 injection monotherapy and in combination with other anti-cancer therapy for advanced malignant tumors of patients. To explore the reasonable dosage of SHR-2002 injection monotherapy and dosage regimen of combination therapy for advanced malignant tumors of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily agrees to participate by giving written informed consent for the study;
2. Male or female aged ≥18 years and ≤70 years at the time of signing the ICF;
3. Histopathologically or cytologically documented advanced or metastatic malignancies;
4. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
5. Life expectancy ≥12 weeks;
6. Adequate organ functions as defined;
7. Female and male patients of reproductive potential must agree to use highly effective contraception during the study treatment period and within 6 months after the last investigational drug administration; Female of childbearing potential must have a negative serum human chorionic gonadotropin (HCG) test within 7 days before the first dose of the investigational drugs and must not be breastfeeding.

Exclusion Criteria:

1. Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis;
2. Patients with active brain metastasis (without medical control or with clinical symptoms), cancerous meningitis, spinal cord compression, or patients with a history of primary tumors of the central nervous system ;
3. Patients with tumor-related pain that cannot be controlled as determined by the investigator;
4. Uncontrollable third-space effusion, such as pleural effusion, pericardial effusion or peritoneal effusion;
5. Systemic anti-tumor therapy within 28 days prior to the first dose of the study treatment;
6. Surgical procedures requiring general anesthesia within 28 days prior to the first dose of the study treatment;
7. Patients who have received >30 Gy of radical radiotherapy within 28 days before the first dose of study treatment;
8. Unresolved CTCAE Grade >1 toxicity attributed to any prior anti-tumor therapy;
9. Use of live attenuated vaccines within 28 days before the first dose of the study treatment;
10. Patients who have received any systemic immunosuppressants within 14 days prior to the first dose of study treatment;
11. Patients with interstitial pneumonitis or interstitial lung disease; past history of interstitial pneumonitis or interstitial lung disease requiring hormone therapy;
12. History of autoimmune diseases;
13. History of clinically significant bleeding symptom or bleeding tendency within 3 months before the first dose of study treatment;
14. History of clinically significant cardiovascular or cerebrovascular diseases within 6 months prior to the first dose of study treatment;
15. Evidence or history of arterial/venous thrombosis within 3 months before the first dose;
16. Prior malignancy (other than current malignant tumor) within 5 ears before the first dose of study treatment;
17. Known history of serious allergic reactions to the investigational product or its main ingredients;
18. History of immunodeficiency;
19. Presence of active hepatitis B or active hepatitis C;
20. Severe infections within 4 weeks prior to the first study treatment;
21. Evidence or history of active pulmonary tuberculosis within 1 year before study entry;
22. any other conditions that are not suitable for participation in the study in the investigator's opinion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | first dose of study medication up to 21 days
  The Maximum tolerated dose of SHR-2002 injection monotherapy or in combination with Camrelizumab for Injection, or SHR-1316 injection, or SHR-1701 injection
Recommended phase II dose | first dose of study medication up to 21 days
  The Recommended phase II dose of SHR-2002 injection monotherapy or in combination with Camrelizumab for Injection, or SHR-1316 injection, or SHR-1701 injection
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | from signature completion of ICF to 90 days after the last dose or to the beginning of the new anti-cancer therapy, whichever came first, assessed up to 24 weeks
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Tmax | 0.5 hour before first dose to the 336 hours after first dose
  PK parameters of single dose of SHR-2002 injection monotherapy
Cmax | 0.5 hour before first dose to the 336 hours after first dose
  PK parameters of single dose of SHR-2002 injection monotherapy
AUC0-t | 0.5 hour before first dose to the 336 hours after first dose
  PK parameters of single dose of SHR-2002 injection monotherapy
AUC0-∞ | 0.5 hour before first dose to the 336 hours after first dose
  PK parameters of single dose of SHR-2002 injection monotherapy
t1/2 | 0.5 hour before first dose to the 336 hours after first dose
  PK parameters of single dose of SHR-2002 injection monotherapy
CL | 0.5 hour before first dose to the 336 hours after first dose
  PK parameters of single dose of SHR-2002 injection monotherapy
Vss | 0.5 hour before first dose to the 336 hours after first dose
  PK parameters of single dose of SHR-2002 injection monotherapy
Cmax, ss | 0.5 hour before second dose to the 30 days after last dose
  PK parameters of multiple doses of SHR-2002 monotherapy
Ctrough, ss | 0.5 hour before second dose to the 30 days after last dose
  PK parameters of multiple doses of SHR-2002 monotherapy
Rac | 0.5 hour before second dose to the 30 days after last dose
  PK parameters of multiple doses of SHR-2002 monotherapy
RO | 0.5 hour before second dose to the 30 days after last dose
  Receptor occupancy, PD indicators of SHR-2002 injection monotherapy
Cytokine concentration | 0.5 hour before second dose to the 30 days after last dose
  PD indicators of SHR-2002 injection monotherapy
Ctrough, ss | 0.5 hour before second dose to the 90 days after last dose
  PK parameters of SHR -2002, Camrelizumab for Injection, SHR-1316 injection and SHR-1701 injection during combination therapy period
Rac | 0.5 hour before second dose to the 90 days after last dose
  PK parameters of SHR -2002, Camrelizumab for Injection, SHR-1316 injection and SHR-1701 injection during combination therapy period
ADA | 0.5 hour before second dose to the 90 days after last dose
  Anti-drug antibody, Immunogenicity of SHR-2002 in monotherapy and combination therapy, Camrelizumab for Injection, SHR-1316 injection and SHR-1701 injection
NAb | 0.5 hour before second dose to the 90 days after last dose
  Immunogenicity of Camrelizumab for Injection, SHR-1316 injection and SHR-1701 injection
ORR | from the date of the first dose to the date of disease progression evaluated based on RECIST v1.1 criteria, death, lost to follow-up, voluntary withdrawal, or initiation of other anti-tumor treatment, whichever occurs first, assessed up to 6 months]
  Objective Response Rate, Efficacy endpoints of SHR-2002 injection monotherapy or in combination with Camrelizumab for Injection, or SHR-1316 injection, or SHR-1701 injection in treatment of patients with Advanced Malignant Tumors
DoR | from the date of the firstly documented tumor response to the date of the firstly documented disease progression or the date of death for any reason, assessed up to 6 months
  Duration of response, Efficacy endpoints of SHR-2002 injection monotherapy or in combination with Camrelizumab for Injection, or SHR-1316 injection, or SHR-1701 injection in treatment of patients with Advanced Malignant Tumors
DCR | from the date of the first dose to the date of the firstly documented disease progression (evaluated based on RECIST v1.1 criteria) or the date of death for any reason, assessed up to 6 months
  Disease control rate, Efficacy endpoints of SHR-2002 injection monotherapy or in combination with Camrelizumab for Injection, or SHR-1316 injection, or SHR-1701 injection in treatment of patients with Advanced Malignant Tumors
PFS | from the date of the first dose to the date of the firstly documented disease progression (evaluated based on RECIST v1.1 criteria) or the date of death for any reason, assessed up to 6 months
  Progression-free survival, Efficacy endpoints of SHR-2002 injection monotherapy or in combination with Camrelizumab for Injection, or SHR-1316 injection, or SHR-1701 injection in treatment of patients with Advanced Malignant Tumors
OS | from the date of the first dose to the date of death for any reason，assessed up to 100 months
  Overall survival, Efficacy endpoints of SHR-2002 injection monotherapy or in combination with Camrelizumab for Injection, or SHR-1316 injection, or SHR-1701 injection in treatment of patients with Advanced Malignant Tumors

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Henan Science and Technology University First Affiliated Hospital, Luoyang, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided